CLINICAL TRIAL: NCT06527820
Title: Aim 2 - Conversations Can Save Lives: TALKing About Buprenorphine & Methadone for Opioid Use Treatment Initiation (TALK ABOUT It)
Brief Title: Aim 2 - Conversations Can Save Lives: TALKing About Buprenorphine & Methadone for Opioid Use Treatment Initiation
Acronym: TalkAboutIt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Schoenfeld, MD, Vice Chair of Research, Department of Emergency Medicine, Baystate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BH-24-001
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use Disorder
Keywords: shared decision-making; decision aid; conversation aid; patient-centered care; addiction; emergency medicine
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Before and after trial. ED patients will be enrolled and followed before and after the intervention is delivered to clinicians. Clinicians at one site will receive the intervention and clinicians at control sites will complete outcome collection without receiving the intervention.
Who Masked: Participant
Masking Description: Participants will receive usual care in all encounters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Talk About It (conversation aid) — "Talk About It" is a conversation aid aimed to increase awareness of options and prompt discussion.

SUMMARY:
The increasing morbidity and mortality of the opioid epidemic has necessitated a reevaluation of current addiction treatment paradigms: medications for opioid use disorder, such as buprenorphine and methadone, are effective in decreasing one's risk of death and disability from opioid use, but are underutilized and often difficult to access. The 5000 Emergency Departments (EDs) in the US are potential additional locales for medication initiation, but currently only a small minority of ED patients with opioid use disorder are started on medications. This study will refine and pilot an intervention called Talk About It which aims to foster patient-centered care, 'meet patients where they are' for addiction treatment, and increase treatment initiation and adherence via facilitating Shared Decision-Making in the ED around these potentially life-saving options.

DETAILED DESCRIPTION:
Participants (ED patients with untreated opioid use disorder) will be enrolled and followed prospectively before and after an ED-wide intervention training clinicians to use "Talk About It," a paper-based conversation aid designed to foster shared decision-making about the decision to start methadone and buprenorphine.

Outcomes will include the initiation of medications, treatment adherence, and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 and older
* presenting with indications for Medications for Opioid Use Disorder (MOUD) initiation (opioid overdose, opioid withdrawal, complications of injection opioid use, untreated OUD)
* not currently on buprenorphine or methadone (in the past 7 days).

(Buprenorphine is FDA approved for patients aged 16 and older, so 16- and 17-year-olds may be included with parental consent.)

Exclusion Criteria:

* No Opioid Use Disorder (OUD)
* already on MOUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of Talk About It (1) | At 18 months
  Clinician report of number of times they utilized the Talk About It Tool in preceding 12 months
Uptake of Talk About It (2) | At 6-18 months
  Number of paper versions of Talk About It tool shared with patients each month as monitored by research staff
Uptake of Talk About It (3) | At 6-18 months
  Number of times the digital version of Talk About It is accessed for clinical care each month (webpage use monitoring software)
Uptake of Talk About It (4) | At 6-18 months
  Number of times patient reports using Talk About It on follow-up survey
Medications for Opioid Use Disorder (MOUD) initiation | From 0-24 months
  1. Rate of Methadone or buprenorphine started in ED (via EHR)
  2. Rate of Prescription written for buprenorphine
Recruitment: Clinician enrollment | From 0-12 months
  Average number of eligible clinicians who complete training and survey instruments
Recruitment: Patient enrollment | From 0-24 months
  Average number of eligible patients who are enrolled each month
Acceptability/Feasibility of Talk About It | At 6 and 18 months
  The Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), Feasibility of Intervention Measure (FIM) scales are brief, validated scales that clinicians will answer regarding acceptability, appropriateness, and feasibility of the intervention. Trained clinicians will complete these scales twice (once immediately after training and once 12 months after training. Range 1-5 with higher meaning better

SECONDARY OUTCOMES:
Knowledge/Awareness | From 0-24 months
  Patients will complete a post-ED knowledge test developed by Steering Committee
Perception of clinicians' compassion | From 0-24 months
  Patients will complete the Sinclair Compassion Questionnaire (SCQ) which assessed their perception of their clinician's compassion (5 questions, range 1-5, higher = better)
Perceived Stigma | From 0-24 months
  Patients will complete a Modified Perceived Stigma of Addiction Scale (PSAS) which assess their perception of their clinician's stigma (Q1 binary, Q2-4, range 1-5 with higher = more stigma)
Attitudes towards methadone | From 0-24 months
  Patients will complete the Attitudes About Methadone (OAM-5) to assess whether the intervention has changed negative attitudes about methadone
Attitudes towards buprenorphine | From 0-24 months
  Patients will complete the Attitudes About Buprenorphine (modified OAM-5) to assess whether the intervention has changed negative attitudes about buprenorphine
Engagement/SDM | From 0-24 months
  Patients will complete the Shared Decision-Making Process Scale (SDM-P) to assess their perceived involvement in decision-making (4 questions, scored 0/1 with higher = more engagement)
Trust | From 0-24 months
  Patients will complete the validated 5-item Trust in Physician Scale to assess their trust in the physician (5 questions, 1-5, with higher = more trust; 1 question reverse coded)
Readiness to change | From 0-24 months
  Patients will fill out the Contemplation ladder scale (1-7), a validated tool to assess readiness for drug abstinence
Stigma | From 0-24 months
  Clinicians will complete the Opening Minds Stigma Scale for Health Care Providers (OMS-HC) twice to assess for changes in stigma (19 questions, each 1-5, lower scrore = less stigma)
Self-efficacy for conversations about MOUD | From 0-24 months
  Clinicians will complete the Self-efficacy in clinical communication scale (SE-12) to assess for changes in self-efficacy around communication (12 questions, response options 1-10, higher score = more self efficacy
Adherence to MOUD | From 0-24 months
  Patients will report their 14- and 30- day use of MOUD, which will be confirmed in the EHR; 60 day adherence will be obtained from EHR and methadone clinics
Illegal opioid use | From 0-24 months
  Patients will report their 14- and 30- day use of illegal opioids

CONTACTS AND LOCATIONS:
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States